CLINICAL TRIAL: NCT05594498
Title: A Pilot Study of StrataXRT in the Prevention of Radiation Dermatitis in Breast Cancer Patients Undergoing Adjuvant Radiotherapy
Brief Title: A Study of StrataXRT in the Prevention of Radiation Dermatitis in Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Edward Chow, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: StrataXRT
Record Dates: First submitted 2022-10-13; First posted 2022-10-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Skin toxicity; StrataXRT; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: All patients will receive the StrataXRT intervention. StrataXRT will be given to patients in one of five patient populations:
  1. Patients with large breasts (minimum of band size of 36 inches or cup size C) treated in the prone position-breast radiation only
  2. Patients with large breasts (minimum of band size of 36 inches or cup size C) treated in the supine position---breast radiation only
  3. Patients with locoregional breast radiation (any breast size)
  4. Patients with local chest wall radiation alone
  5. Patients with locoregional chest wall radiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- StrataXRT Arm (Experimental): This is a single-arm trial where all patients will receive the intervention of StrataXRT.
  Interventions: Device: StrataXRT

INTERVENTIONS:
Device: StrataXRT — StrataXRT is a silicone-based film-forming topical gel that may help in reducing radiation dermatitis.

SUMMARY:
For breast cancer patients undergoing adjuvant radiotherapy, radiation dermatitis (RD) is a common occurrence that can negatively impact patients' quality of life (QOL). RD often presents as erythema, pruritus, and/or edema and in more severe cases, skin breakage can occur, resulting in moist desquamation. StrataXRT is a silicone-based film-forming topical gel. Recent studies have shown the benefits of StrataXRT, but with mixed results. A recent randomized controlled trial published in 2022 found that in breast cancer patients (n=100), the use of StrataXRT significantly reduced the mean size of the radiation-induced dermatitis area (p=0.002) when compared to the control group. Additionally, another study (n=49) demonstrated significant differences in the Erythema Index (EI) (p=0.001) and Melanin Index (MI) (p=0.005) between StrataXRT compared to the use of Xderm, a moisturizer cream. To validate the finding of the previous studies a pilot study testing the efficacy of StrataXRT has been proposed. In this study, 50 patients will use Strata XRT on their breast/chest wall during radiation treatment. Their skin will be assessed throughout and post-treatment. Investigators hypothesize the severity of skin reactions will be less for patients using Strata XRT when compared to historical data from our centre.

DETAILED DESCRIPTION:
For breast cancer patients undergoing adjuvant radiotherapy, radiation dermatitis (RD) is a common occurrence that can negatively impact patients' quality of life (QOL). RD often presents as erythema, pruritus, and/or edema and in more severe cases, skin breakage can occur, resulting in moist desquamation. StrataXRT is a silicone-based film-forming topical gel, intended to be self-applied by the patients. As a result of the product's film-forming property, the gel can also be applied to the axilla and supraclavicular area. Due to the more versatile method of application, it is also possible that this product would be feasible for patients with large breasts, and patients treated in the prone position. This gel has the potential to reduce RD in patients with large breasts and patients receiving regional radiation.

StrataXRT has been shown to be non-inferior to Mepitel Film, a silicone dressing, in the prevention of RD. A study compared the rates of moist desquamation and CTCAE scoring in 44 breast cancer patients. Half the breast was covered with Mepitel Film and the other half with StrataXRT. The results showed no significant differences in the rate of moist desquamation or severity of RD assessed on the CTCAE between groups. There have been two randomized control trials conducted that showed promising results using StrataXRT. One of the studies found that in breast cancer patients (n=100), the use of StrataXRT significantly reduced the mean size of the radiation-induced dermatitis area (p=0.002) when compared to the control group. Additionally, RD as scored by the CTCAE was found to be significantly more severe in the control group. Another randomized control trial (n=49) demonstrated significant differences in the Erythema Index (EI) (p=0.001) and Melanin Index (MI) (p=0.005) between StrataXRT compared to the use of Xderm, a moisturizer cream. The EI and MI are alternative methods of measuring RD, using electrochemical reflectance most often with a handheld spectrophotometer.

There is limited research available on the ability of StrataXRT to prevent RD, and the available research presents major limitations and variability across studies. Measurement tools are inconsistent, and even when the scales are the same across studies, there is significant variability in the results. Further StrataXRT has not been widely adopted in North America for the prevention of RD. Therefore to validate the efficacy of StrataXRT in the prevention of severe radiation dermatitis a feasibility study using five patient populations will be conducted:

1. Patients with large breasts (minimum of band size of 36 inches or cup size C) treated in the prone position-breast radiation only
2. Patients with large breasts (minimum of band size of 36 inches or cup size C) treated in the supine position---breast radiation only
3. Patients with locoregional breast radiation (any breast size)
4. Patients with local chest wall radiation alone
5. Patients with locoregional chest wall radiation

The results of the feasibility study can go on to guide the development of a large multi-center randomized controlled trial to further validate the use of StrataXRT and potentially increase the adoption rate in North America.

The primary objective is to evaluate the feasibility of StrataXRT in the prevention of RD. Secondary objectives will include patient- and clinician-reported skin reactions and the presence of moist desquamation with the use of StrataXRT. As well as patient QOL and patient and clinician satisfaction with StrataXRT.

Patients will be approached by clinical research assistants (CRA) at their planning appointment. Here the CRA will introduce the study and provide them with an information sheet to read. After all information has been reviewed if patients are interested the CRA will obtain consent. All patients will receive StrataXRT to use during their treatment. Radiation treatment will be delivered as prescribed by the treating radiation oncologist. A trained CRA will teach the patients how to apply the StrataXRT on their first day of treatment. The CRA will make sure the patients know how and where to apply the gel. Patients will be asked to self-apply the StrataXRT at least twice daily and record how many times a day they apply it using a diary given to them on their first day.

Once a week during patients' regular visits with their treating radiation oncologist, patients and clinicians will be asked to complete assessments. On the first and last day of treatment, a photo of the patient's breasts/chest wall will be taken. At their last treatment, they will also be asked to complete additional assessments.

After completing radiation treatment, patients will be called for the following 6 weeks to complete assessments. Patients will be asked to return for an in-person assessment for their 2-week follow-up, instead of a telephone follow-up. A photo of the breasts/chest wall will be taken at this appointment and both patients and clinicians will be asked to complete assessments. A telephone follow-up will also take place 6-months post radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histological confirmation of breast malignancy (invasive or in situ carcinoma) or phyllodes
* Patient are scheduled to receive conventionally - (50 Gy/25) or hypofractionated (40 Gy/15 or 42.6 Gy/16)
* Can communicate in English or be aided by a translator

Exclusion Criteria:

* Patient had previous radiation therapy to the treatment area
* Patient will receive partial breast external beam radiation or brachytherapy
* Patients scheduled to receive extreme hypofractionation (26 Gy/ 5)
* Patients with active rash, pre-existing dermatitis, or other conditions within the treatment area that may make skin assessment for the study difficult per treating physician discretion.
* Patients with known allergy or sensitivity to silicone
* Concomitant cytotoxic chemotherapy
* Bilateral breast pathology requiring concurrent bilateral breast radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinician grading of acute skin toxicity | Within 3-months following radiation treatment
  Measured by the Common Terminology Criteria for Adverse Events; graded on a scale from 0 (best) to 4 (worst) assessed by clinicians

SECONDARY OUTCOMES:
Patient reports of acute toxicity | Within 3-months following radiation treatment
  Measured by the Skin Symptom Assessment; items include itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling, and trouble fitting brassieres graded on a four-point scale using "not at all", "a little", "quite a bit", or "very much"
Clinicians reports of acute toxicity | Within 3-months following radiation treatment
  Measured by the Skin Symptom Assessment; items include itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling, and trouble fitting brassieres graded on a four-point scale using "not at all", "a little", "quite a bit", or "very much"
Incidence of moist desquamation | Within 3-months following radiation treatment
  Measured using a yes/no answered by clinicians
Degree of acute skin toxicity and interference with daily functioning | Within 3-months following radiation treatment
  Measured by the Radiation Induced Skin Reaction Assessment System; researcher subscales for erythema and dry desquamation rated from 0 (best) to 4 (worst); researcher subscale for moist desquamation rated from 0 (best) to 6 (worst); researcher subscale for necrosis rated from 0 (best) to 10 (worst); patient subscales for tenderness/discomfort/pain, itchiness, burning sensation, and interference with daily activities rated from 0 (best) to 3 (worst).
Observable differences between treated and non-treated breasts/chest wall | Within 3-months following radiation treatment
  Determined by photographs of the treated and non-treated breast/chest wall
Patient-reported quality of life | Within 3-months following radiation treatment
  Measured using the Skindex-16; measures if 16 different symptoms have bothered the patient on a scale of 0 to 6 (0=never bothered, 6=always bothered).
Patient satisfaction with StrataXRT | Within 3-months following radiation treatment
  Measured using a patient satisfaction questionnaire
Clinician satisfaction with StrataXRT | Within 3-months following radiation treatment
  Measured using a constructed clinician satisfaction questionnaire
Cost analysis of StrataXRT | Within 3-months following radiation treatment
  Measured using records of use of StrataXRT for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Edward LW Chow, MBBS, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ahn S, Sung K, Kim HJ, Choi YE, Lee YK, Kim JS, Lee SK, Roh JY. Reducing Radiation Dermatitis Using a Film-forming Silicone Gel During Breast Radiotherapy: A Pilot Randomized-controlled Trial. In Vivo. 2020 Jan-Feb;34(1):413-422. doi: 10.21873/invivo.11790. PMID 31882508
- [Derived] Kuszaj O, Day M, Zhang L, Wong H, Lee SF, Kwan JYY, Wang AJ, Bayrakdarian S, Karam I, Tran W, Chow E. Validation of the Skin Symptom Assessment (SSA) questionnaire for the evaluation of radiation dermatitis in breast cancer patients. Support Care Cancer. 2024 Sep 24;32(10):683. doi: 10.1007/s00520-024-08890-9. PMID 39316164
- [Derived] Kennedy SKF, Gojsevic M, Rajeswaran T, Zhang L, Kuszaj O, Day M, Karam I, Vesprini D, Leung E, Szumacher E, Rakovitch E, Soliman H, Chen H, Lee SF, Behroozian T, Tran W, Wronski M, Gallant F, Carothers K, Yewhans T, Wong C, Wong H, Chow E. StrataXRT for the prevention of acute radiation dermatitis in breast cancer: a pilot study. Support Care Cancer. 2024 Sep 18;32(10):670. doi: 10.1007/s00520-024-08851-2. PMID 39292351
- See also: StrataXRT is non-inferior to Mepitel Film — https://www.postersessiononline.eu/173580348_eu/congresos/ESTRO38/aula/-EP_1286_ESTRO38.pdf
- See also: The Investigation of Prophylactic Effect of StrataXRT Gel on Radiation-Induced Dermatitis in Breast Cancer Patients: A Randomized Clinical Trial — https://dx.doi.org/10.30476/mejc.2021.86775.1372